CLINICAL TRIAL: NCT03178396
Title: Effects and Mechanisms of Melatonin on Blood Pressure, Insulin Resistance, and Platelets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15F.572; R01HL096593 (NIH)
Record Dates: First submitted 2017-05-26; First posted 2017-06-06 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Prehypertension; Healthy
MeSH Terms: conditions — Prehypertension | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Young, intervention (Experimental): patients ages 18-45, taking melatonin
  Interventions: Dietary Supplement: melatonin
- Young, control (No Intervention): patients ages 18-45, usual care
- Older, intervention (Experimental): patients ages 60 and older, taking melatonin
  Interventions: Dietary Supplement: melatonin
- Older, control (No Intervention): patients ages 60 and older, usual care

INTERVENTIONS:
Dietary Supplement: melatonin — controlled release, 9 mg taken 30 minutes before bedtime x 6 weeks
  Other Names: Life Extension Foundation
  Arms: Older, intervention; Young, intervention

SUMMARY:
The investigators will be studying the effect of melatonin on blood pressure, insulin resistance, and platelets, along with possible reasons for how melatonin cases these effects.

DETAILED DESCRIPTION:
The investigators will be studying the effect of melatonin on blood pressure and insulin resistance, and possible reasons for how melatonin works on blood pressure and IR. Along with blood testing to measure adipokines, insulin resistance (IR), and platelet function (how well your blood clots), 24-hour ambulatory blood pressure monitoring (ABPM) will be used to measure blood pressure, since ABPM is the gold standard (best method) for accurate assessment of blood pressure status and associated cardiovascular risk. Vascular (blood vessel) function, IR, adipokine levels and sleep quality will also be measured. All study endpoints will be measured at baseline and following 6 weeks of daily melatonin 9 mg dosing.

ELIGIBILITY:
Inclusion Criteria:

* Normotensive (SBP <120) or prehypertensive (SBP = 120-139 mm Hg)
* Age: Young/middle-aged (ages 18-45) and (2) 10 elderly subjects ages 65 and older

Exclusion Criteria:

* Patients with a diagnosis of

  * clinical hypertension and/or diabetes mellitus
  * pregnancy
  * coronary or cerebrovascular disease
  * collagen vascular disease,
  * organ failure (heart, kidney, liver).
* Patients taking anti-inflammatory medications: NSAIDs, corticosteroids, thiazolidinediones, and statins,
* Patients who have taken melatonin previously in the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2016-08-09 (Actual); Study Completion 2016-08-09 (Actual)

PRIMARY OUTCOMES:
Office Systolic Blood pressure change | Baseline to 6 weeks
  Change in Systolic blood pressure measured in the office at 6 weeks
Office Diastolic Blood pressure change | Baseline to 6 weeks
  Change in Diastolic blood pressure measured in the office at 6 weeks
Ambulatory Systolic Blood pressure change | Baseline to 6 weeks
  Change in 24 hour average Systolic blood pressure at 6 weeks
Ambulatory Diastolic Blood pressure change | Baseline to 6 weeks
  Change in 24 hour average Diastolic blood pressure at 6 weeks
HOMA: Homeostasis Model Assessment change | Baseline to 6 weeks
  Insulin sensitivity measure change at 6 weeks
QUICKI: Quantitative insulin sensitivity check index change | Baseline to 6 weeks
  Insulin sensitivity measure change at 6 weeks

SECONDARY OUTCOMES:
Arachidonic acid stimulated aggregation change | Baseline to 6 weeks
  Platelet activity measure change at 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Cheng, MD,PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Summarized data, available immediately by contacting PI